CLINICAL TRIAL: NCT01863849
Title: Tolerability and Immunogenicity Study of Fluval AB Suspension for Injection (Trivalent, Seasonal Influenza Vaccine, Active Ingredient Content: 15 μgHA/Strain/0.5mL) for the Use in the Season 2013/2014 in Adult and Elderly Subjects
Brief Title: Tolerability and Immunogenicity Study of Fluval AB Suspension for Injection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fluart Innovative Vaccine Ltd, Hungary (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FluvalAB-H-YL2013
Record Dates: First submitted 2013-05-23; First posted 2013-05-29 (Estimated); Results first posted 2021-04-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-03

CONDITIONS: Influenza Prophylaxis
Keywords: uncontrolled; open; multi-centre; immunogenicity and tolerability; two groups according to age (18-59 years and ≥60 years)
MeSH Terms: interventions — Vaccination; Injections

STUDY DESIGN:
Intervention Model Description: parallel-group, in two age groups
Oversight: Data Monitoring Committee: No

ARMS (2):
- Age group 1: adults (18-59 years) (Experimental): Intervention: Vaccination with Fluval AB suspension for injection.
  Dosage: A single dose (0.5 ml) vaccine, administered intramuscularly.
  Interventions: Biological: Vaccination with Fluval AB suspension for injection
- Age group 2: elderly (> 60 years) (Experimental): Intervention: Vaccination with Fluval AB suspension for injection.
  Dosage: A single dose (0.5 ml) vaccine, administered intramuscularly.
  Interventions: Biological: Vaccination with Fluval AB suspension for injection

INTERVENTIONS:
Biological: Vaccination with Fluval AB suspension for injection — Single intramuscular injection with Fluval AB suspension for injection in both age groups

SUMMARY:
To assess immunogenicity of a single intramuscular injection of Fluval AB suspension for injection (trivalent, seasonal influenza vaccine, active ingredient content: 15 μgHA/0.5mL of seasonal A/H1N1, A/H3N2 and B influenza antigens each), as measured by haemagglutination inhibition (HI) test.

DETAILED DESCRIPTION:
Aim of the study:

To assess immunogenicity and safety of Fluval AB seasonal influenza vaccine with 3 x 15 μgHA active ingredient in two age groups (18-59 years and ≥60 years) in accordance with CPMP/BWP/214/96: "Note for Guidance on Harmonization of Requirements for Influenza Vaccines", 12 March 1997

Primary objective:

To assess immunogenicity of a single intramuscular injection of Fluval AB suspension for injection (trivalent, seasonal influenza vaccine, active ingredient content: 15 μgHA/0.5mL of seasonal A/H1N1, A/H3N2 and B influenza antigens each), as measured by haemagglutination inhibition test.

Methods:

In this open label, uncontrolled, multi-centre immunogenicity and tolerability study subjects were enrolled in two groups according to age (18-59 years and ≥60 years) and assigned to the following vaccine group:

Group 1: Single injection of Fluval AB suspension for injection. Subjects were observed for 30 minutes after the injection on Visit 1 (Day 0) for any immediate reactions.

All subjects were requested to complete a diary card to record local reactions (injection site pain, erythema, swelling, induration and ecchymosis) and systemic reactions (fever, shivering, headache, malaise, fatigue, sweating, nausea, myalgia and arthralgia) started on the day of vaccination on Visit 1 (Day 0) until 7 (seven) days following that.

All adverse events were collected during the period of Visit 1 (Day 0) to Visit 2 (between Day 21 and Day 28).

Serum samples for immunogenicity assays were collected immediately before immunization on Visit 1 (Day 0) and on Visit 2 (between Day 21 and Day 28) in all subjects. Immunogenicity was evaluated by HI test.

ELIGIBILITY:
Inclusion Criteria:

* Adult persons aged 18 to 59 years, elderly persons aged ≥60 years from both sexes, mentally competent;
* Are in good health (as determined by vital signs and existing medical condition) or are in stable medical condition. Subjects will not be excluded with known adequately treated clinically significant organ or systemic diseases (e.g. asthma or diabetes), such that, in the opinion of the investigator, the significance of the disease will not compromise the subject's participation in the study;
* Female volunteers aged 18-59 years (i.e. participants of childbearing potential) with a negative result from the urine pregnancy test prior to vaccination who agrees to use an acceptable contraception method or abstinence throughout the trial and not become pregnant for the duration of the study;
* Capability of participants to understand and comply with planned study procedures;
* Participants provide written Informed Consent (IC) prior to initiation of study procedures;
* Absence of existence of any exclusion criteria.

Exclusion Criteria:

* Pregnancy, breast feeding or positive urine pregnancy test at baseline prior to vaccination. Female subjects who are able to bear children but not willing to use an acceptable contraception method for the duration of the study.
* Known hypersensitivity to eggs, chicken protein, thiomersal, formaldehyde, gentamycin, ciprofloxacin, neomycin, vancomycin or any other component of the vaccine;
* History of Guillain-Barré syndrome;
* History of neurological symptoms or signs, or anaphylactic shock following administration of any vaccine;
* Serious disease, such as cancer, autoimmune disease, advanced arteriosclerotic disease, complicated diabetes mellitus, acute or progressive hepatic disease, acute or progressive renal disease, congestive heart failure;
* Immunosuppressive therapy within 36 months prior to vaccination;
* Concomitant corticosteroid therapy, including high-dose inhaled corticosteroids;
* Receipt of immunostimulants;
* Receipt of parenteral immunoglobulin, blood products and/or plasma derivate within 3 months prior to vaccination;
* Suspected or known HIV, HBV or HCV infection;
* Acute disease and/or axillary temperature ≥37oC within 3 days prior to vaccination;
* Vaccine therapy within 4 weeks prior to vaccination;
* Influenza vaccination (any kind) within 6 months prior to vaccination;
* Experimental drug therapy within 4 weeks prior to vaccination;
* Concomitant participation in another clinical study;
* Any condition which, in the opinion of the investigator, may interfere with the evaluation of the study;
* Past or current psychiatric disease of the volunteer that upon judgement of the investigator may have effect on the objective decision-making of the volunteer;
* Alcohol or drug abuse of the participant.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-08-22; Primary Completion 2013-09-17 (Actual); Study Completion 2013-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zsolt Németh, Study Chair — Fluart Innovative Vaccines Ltd.
Locations (3):
- Hungary (3):
  - Family Doctor's Office, Budapest
  - District Doctor's Office, Pilisvörösvár
  - District Doctor's Office, Szentendre

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Age Group 1: Adults (18-59 Years); Age Group 2: Elderly (> 60 Years): Intervention: Vaccination with Fluval AB suspension for injection.
  Dosage: A single dose (0.5 ml) vaccine, administered intramuscularly.
  Vaccination with Fluval AB suspension for injection: Single intramuscular injection with Fluval AB suspension for injection in both age groups
Period: Overall Study
Arm/Group | Age Group 1: Adults (18-59 Years) | Age Group 2: Elderly (> 60 Years)
Started | 60 | 60
Completed | 59 | 60
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Primary analysis is conducted on the PP population.
Groups:
- Age Group 2: Elderly (>60 Years): Intervention: Vaccination with Fluval AB suspension for injection.
  Dosage: A single dose (0.5 ml) vaccine, administered intramuscularly.
- Total: Total of all reporting groups
Arm/Group | Age Group 1: Adults (18-59 Years) | Age Group 2: Elderly (>60 Years) | Total
Number analyzed (Participants) | 59 | 60 | 119
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 59 | 16 | 75
  >=65 years | 0 | 44 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (9.69) | 69.8 (6.87) | 58.1 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 31 | 68
  Male | 22 | 29 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 59 | 60 | 119
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Hungary | 59 | 60 | 119

OUTCOME MEASURES:

1. Primary Outcome: Change in Geometric Mean Titre Ratio, A/H1N1 Strain
Description: Ratio of Day 0 and Day 21-28 antihaemagglutination inhibition titres
  Requirement (Age group 1): ≥ 2.5 Requirement (Age group 2): ≥ 2.0
Time Frame: 21-28 days after vaccination
Population: PP population (subjects whose antihaemagglutination inhibition titres are available both Day 0 and Day 21-28 visits)
Measure: Mean (95% Confidence Interval); unit: Ratio of Day 0 and Day 21-28 titres
Arm/Group | Age Group 1: Adults (18-59 Years) | Age Group 2: Elderly (>60 Years)
Number analyzed (Participants) | 59 | 60
Ratio of Day 0 and Day 21-28 titres | 3.13 [2.63 to 3.72] | 3.17 [2.65 to 3.8]

2. Primary Outcome: Change in Geometric Mean Titre Ratio, A/H3N2 Strain
Description: as for outcome 1
Time Frame: 21-28 days after vaccination
Population: PP population (subjects whose antihaemagglutination inhibition titres are available both Day 0 and Day 21-28 visits)
Measure: Mean (95% Confidence Interval); unit: Ratio of Day 0 and Day 21-28 titres
Arm/Group | Age Group 1: Adults (18-59 Years) | Age Group 2: Elderly (> 60 Years)
Number analyzed (Participants) | 59 | 60
Ratio of Day 0 and Day 21-28 titres | 3.58 [2.92 to 4.38] | 3.86 [3.19 to 4.68]

3. Primary Outcome: Change in Geometric Mean Titre Ratio, B Strain
Description: as for outcome 1
Time Frame: 21-28 days after vaccination
Population: PP population (subjects whose antihaemagglutination inhibition titres are available both Day 0 and Day 21-28 visits)
Measure: Mean (95% Confidence Interval); unit: Ratio of Day 0 and Day 21-28 titres
Arm/Group | Age Group 1: Adults (18-59 Years) | Age Group 2: Elderly (> 60 Years)
Number analyzed (Participants) | 59 | 60
Ratio of Day 0 and Day 21-28 titres | 3.58 [2.96 to 4.32] | 4.29 [3.45 to 5.33]

4. Primary Outcome: Seroconversion, A/H1N1 Strain
Description: Percentage of subjects seroconverted or had a significant increase in titres
  Requirement (Age group 1): > 40 % Requirement (Age group 2): > 30 %
Time Frame: 21-28 days after vaccination
Population: PP population (subjects whose antihaemagglutination inhibition titres are available both Day 0 and Day 21-28 visits)
Measure: Number; unit: percentage of subjects seroconverted
Arm/Group | Age Group 1: Adults (18-59 Years) | Age Group 2: Elderly (> 60 Years)
Number analyzed (Participants) | 59 | 60
percentage of subjects seroconverted | 59.3 | 66.7

5. Primary Outcome: Seroconversion, A/H3N2 Strain
Description: as for outcome 4
Time Frame: 21-28 days after vaccination
Population: PP population (subjects whose antihaemagglutination inhibition titres are available both Day 0 and Day 21-28
Measure: Number; unit: percentage of subjects seroconverted
Arm/Group | Age Group 1: Adults (18-59 Years) | Age Group 2: Elderly (> 60 Years)
Number analyzed (Participants) | 59 | 60
percentage of subjects seroconverted | 69.5 | 70.0

6. Primary Outcome: Seroconversion, B Strain
Description: as for outcome 4
Time Frame: 21-28 days after vaccination
Population: PP population (subjects whose antihaemagglutination inhibition titres are available both Day 0 and Day 21-28
Measure: Number; unit: percentage of subjects seroconverted
Arm/Group | Age Group 1: Adults (18-59 Years) | Age Group 2: Elderly (> 60 Years)
Number analyzed (Participants) | 59 | 60
percentage of subjects seroconverted | 54.2 | 65.0

7. Primary Outcome: Seroprotection, A/H1N1 Strain
Description: Percentage of subjects seroprotected
  Requirement (Age group 1): > 70 % Requirement (Age group 2): > 60 %
Time Frame: 21-28 days after vaccination
Population: PP population (subjects whose antihaemagglutination inhibition titres are available both Day 0 and Day 21-28 visits)
Measure: Number; unit: percentage of subjects seroprotected
Arm/Group | Age Group 1: Adults (18-59 Years) | Age Group 2: Elderly (> 60 Years)
Number analyzed (Participants) | 59 | 60
percentage of subjects seroprotected | 94.9 | 96.7

8. Primary Outcome: Seroprotection, A/H3N2 Strain
Description: Percentage of subjects seroprotected
  Requirement (Age group 1): > 70 % Requirement (Age group 2): > 60 %
Time Frame: 21-28 days after vaccination
Population: PP population (subjects whose antihaemagglutination inhibition titres are available both Day 0 and Day 21-28 visits)
Measure: Number; unit: percentage of subjects seroprotected
Arm/Group | Age Group 1: Adults (18-59 Years) | Age Group 2: Elderly (> 60 Years)
Number analyzed (Participants) | 59 | 60
percentage of subjects seroprotected | 100.0 | 100.0

9. Primary Outcome: Seroprotection, B Strain
Description: Percentage of subjects seroprotected
  Requirement (Age group 1): > 70 % Requirement (Age group 2): > 60 %
Time Frame: 21-28 days after vaccination
Population: PP population (subjects whose antihaemagglutination inhibition titres are available both Day 0 and Day 21-28 visits)
Measure: Number; unit: percentage of subjects seroprotected
Arm/Group | Age Group 1: Adults (18-59 Years) | Age Group 2: Elderly (> 60 Years)
Number analyzed (Participants) | 59 | 60
percentage of subjects seroprotected | 79.7 | 78.3

ADVERSE EVENTS:
Time Frame: 21-28 days after vaccination
Description: Subjects were observed for 30 minutes after the injection on Visit 1 (Day 0) for any immediate reactions.
  All subjects were requested to complete a diary card to record local and systemic reactions started on the day of vaccination on Visit 1 (Day 0) until 7 (seven) days following that.
  All adverse events were collected during the period of Visit 1 (Day 0) to Visit 2 (between Day 21 and Day 28).
Arm/Group | Age Group 1: Adults (18-59 Years) | Age Group 2: Elderly (> 60 Years)
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/60
Other Adverse Events (participants affected / at risk) | 51/59 | 14/60
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Age Group 1: Adults (18-59 Years) (N=59) | Age Group 2: Elderly (> 60 Years) (N=60)
vaccination site pain (General disorders) | 19 (19) | 4 (4) — pain at vaccination site
vaccination site swelling (General disorders) | 9 (9) | 5 (5) — swelling at vaccination site
vaccination site erythema (General disorders) | 13 (13) | 3 (3) — erythema at vaccination site
vaccination site induration (General disorders) | 11 (11) | 1 (1) — induration at vaccination site
pyrexia (Gastrointestinal disorders) | 2 (2) | 0 (0) — fever
headache (Nervous system disorders) | 7 (7) | 1 (1)
malaise (General disorders) | 2 (2) | 2 (2)
hyperhidrosis (General disorders) | 0 (0) | 1 (1) — sweat
myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) — muscle pain
arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — joint pain
vaccination site haematoma (General disorders) | 2 (2) | 0 (0) — haematoma at vaccination site

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that the sponsor in the frames of the general confidentiality agreement is that the PI cannot release any information concerning the study without the prior consent of the sponsor. To further specification is provided.